CLINICAL TRIAL: NCT03237546
Title: The Use of Serratus Block for Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-00070
Record Dates: First submitted 2017-07-31; First posted 2017-08-02 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Cardiac Surgery
Keywords: Robotic Cardiac Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Serratus blocks (Active Comparator): The serratus plane is interstitial tissue, below the serratus muscle. The injection of bupivacaine numbs the anterior branch of the thoracodorsal nerve. This technique allows for the medication to diffuse along the area of the serratus plane to provide numbing of that area. Upon completion of the block, the patient will be evaluated for extubation and emerged from general anesthesia if appropriate.
  Interventions: Procedure: Anesthetic regimen including SB
- PCA-alone (no block) (Active Comparator): All subjects will receive fentanyl intravenous patient controlled anesthesia pumps as part of standard care. The amount of fentanyl self-administered by the patient or given by a clinician during 24 hours following surgery will be compared amongst the two groups.
  Interventions: Procedure: Anesthetic regimen including SB or no block

INTERVENTIONS:
Procedure: Anesthetic regimen including SB — Group receiving general anesthesia with the serratus block
  Arms: Serratus blocks
Procedure: Anesthetic regimen including SB or no block — Group receiving general anesthesia alone
  Arms: PCA-alone (no block)

SUMMARY:
The purpose of this randomized, un-blinded study is to determine if serratus blocks or Patient Controlled Analgesia (PCA)-alone (no block) offer patients adequate pain relief. This study will compare two standard of care pain management options and the patients narcotic requirements in the immediate postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 years of age undergoing robotic cardiac surgery.

Exclusion Criteria:

* Patients who are not candidates for serratus block

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2017-11-13 (Actual); Study Completion 2017-11-13 (Actual)

PRIMARY OUTCOMES:
Amount of intravenous opiates used during the immediate postoperative period | 24 Hours
  The primary endpoint of the study will be comparison of the amount of intravenous opiates used during the immediate postoperative period between the 2 groups, the group receiving general anesthesia with the serratus block and the group receiving general anesthesia alone.

CONTACTS AND LOCATIONS:
Overall Officials: Jennie Ngai, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided